CLINICAL TRIAL: NCT07046533
Title: Evaluation of the Success Rate of Full Coronal Pulpotomy as Compared to Conventional Root Canal Therapy in the Management of Mature First Permanent Molars With Irreversible Pulpitis in Children
Brief Title: Evaluation of the Success Rate of Pulpotomy Versus to Root Canal Therapy in Management of Mature First Permanent Molars With Irreversible Pulpitis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lamiaa Saeed Ahmed Elshiekh (Other)
Responsible Party: Sponsor-Investigator, Lamiaa Saeed Ahmed Elshiekh, Assistant Lecturer of Pediatric Dentistry, Faculty of Dentistry October 6th University, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Cairo2007
Record Dates: First submitted 2025-06-13; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Irreversible Pulpitis (Toothache); Dental Caries (Diagnosis)
Keywords: randomized control trial; vital pulp therapy
MeSH Terms: conditions — Toothache; Dental Caries; Disease | interventions — Pulpotomy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- root canal treatment (Active Comparator): invasive technique depends on removal of all pulp tissue coronal and radicular and restore it with a gutta perch with bioceramic sealer
  Interventions: Procedure: (pulpotomy); Procedure: root canal treatment
- pulpotomy (Experimental): non invasive technique depends on removal of only coronal pulp tissue and restore it with a new material bio c repair
  Interventions: Procedure: (pulpotomy); Procedure: root canal treatment

INTERVENTIONS:
Procedure: (pulpotomy) — non invasive technique depends on remove only the coronal pulp tissue instead of remove all pulp tissue
  Other Names: vital pulp therapy
Procedure: root canal treatment — invasive technique depends on remove all radicular and coronal pulp tissue

SUMMARY:
The goal of This current study compare the clinical & radiographic success rate between two different modalities conventional RCT and VPT using Bio-C-Repair as a pulp capping material to treat young patients with mature first permanent molars with irreversible pulpitis.

DETAILED DESCRIPTION:
The teeth were anesthetized with 4% articaine with adrenaline 1/100,000 , isolated under rubber dam , and sterilized using a cotton pellet soaked in 2.5% sodium hypochlorite (NaOCl). Then carious leisons were removed by using a fresh sterile high-speed diamond bur under copious water irrigation. Upon pulp exposed, the cavity was rinsed with 2.5% NaOCl. The other steps of the treatment proceeded accordingly:

The procedure FP involved the removal of all coronal pulp tissue to the canals orifices level through a fresh sterile high-speed diamond bur Hemostasis was accomplished by compressing a cotton pellet soaked in 2.5% NaOCl over the radicular pulp tissue for 5 min. Then, irrigation with amount of sterile 0.9% sodium chloride (NaCl) solution was gently conducted. Once hemostasis was achieved, the radicular pulp tissue was observed as uniformly reddish pink color. Subsequently, a new type of premixed pulp-capping bio c repair ) was prepared according to the manufacturer's instructions, and a 4-mm layer was directly adapted over the radicular pulp tissue, ensuring that there was not any excess materials on the pulp chamber walls. The access cavity was restored with a liner)and composite restoration all completed in a single visit. Then postoperative radiographs were taken.

RCT was conducted in single visit the pulp tissues were removed from all the root canals, identifying and enlarging canal orifices via fanta Gold rotary , determing the working length with an apex locator. The root canals preparation was conducted by rotary nickel-titanium files, irrigated by using 2.5% NaOCl and 17% ethylenediaminetetraacetic acid (EDTA), and disinfected by using Ca(OH)2.

obturation was performed with gutta-percha and biocermaic sealer, using single cone technique.The access cavity was restored with a liner and resin composite restoration during the same appointment while using rubber dam isolation.

ELIGIBILITY:
Inclusion Criteria:

1. Molars teeth with a history of spontaneous radiating pain indicated IP
2. the pain triggered by hot/cold fluids lasted for several minutes after removing of the stimulus.
3. Molars teeth with no prominent radiolucency at the periapical or furcation regions

Exclusion Criteria:

1. Teeth with continuous bleeding
2. necrosis
3. Teeth could not be restored with direct restoration. Teeth having localized/generalized periodontal diseases (probing pocket depth more than 3 mm).

Teeth with crack fracture. Teeth with internal/external root resorption. Teeth with pulp chamber/canal calcification

Ages: 9 Months to 14 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
success rate | 12 months
  clinically and radiographically success rate according to success criteria